CLINICAL TRIAL: NCT02210845
Title: Impact of Two Lifestyle Strategies for Improving Diabetes Related Health Outcomes in a Specialty Care Setting: A Randomized Controlled Trial
Brief Title: Lifestyle Strategies for Improving Diabetes Outcomes
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tom Elliott (Network)
Responsible Party: Sponsor-Investigator, Tom Elliott, Clinical Associate Professor, BCDiabetes.Ca
Organization: BCDiabetes.Ca (Network)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: DOS-23
Record Dates: First submitted 2014-08-04; First posted 2014-08-07 (Estimated); Last update posted 2017-02-20 (Actual); Status verified 2017-02

CONDITIONS: Diabetes
Keywords: Diabetes; Supervised Exercise; Weight loss
MeSH Terms: conditions — Diabetes Mellitus; Weight Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Financially incentivized weight loss (Active Comparator): Participants can be assigned to the financially incentivized weight loss group in which they can receive 50 dollars at the end of the month if they achieve their monthly weight loss goal.
  Interventions: Behavioral: Financially incentivized weight Loss
- Standard of Care (Placebo Comparator): Participants can be assigned to standard of care where they receive no intervention.
  Interventions: Other: Standard Care at BCDiabetes
- Supervised Exercise (Active Comparator): Participants can be assigned to the supervised exercise arm which they will receive supervised professional training once a week.
  Interventions: Behavioral: Supervised exercise

INTERVENTIONS:
Behavioral: Supervised exercise — Supervised exercise intervention is training with professional trainers once a week. It will include aerobic exercise tailored to the individual participant.
  Arms: Supervised Exercise
Behavioral: Financially incentivized weight Loss — Financially incentivized weight loss encourages participants to achieve a monthly goal weight reduction for a 50 dollars prize.
  Arms: Financially incentivized weight loss
Other: Standard Care at BCDiabetes — usual care dictated by GCP at BCDiabetes.ca
  Arms: Standard of Care

SUMMARY:
The objective of this study is to investigate whether a behavioral modification intervention in the form of either a 6-month supervised training program or a 6-month financial incentive weight loss program, results in improvement of diabetes outcome such as overall sugar control and lipid control.

DETAILED DESCRIPTION:
This is a single-center, prospective, unblinded, randomized, controlled, clinical trial of 200 subjects randomized to either a Supervised Training Program (STP), Incentivized Weight Loss (IWL) or Standard of Care (SoC).

Subjects randomized to the SoC group will be asked to return for regular 3-monthly clinic visits and for diet and exercise recommendations.The STP group will be offered once-weekly one hour supervised training sessions at no charge for a period of six months in the bcdiabetes.ca fitness center (located in the Vancouver General Hospital Employee Centre gym).

The IWL group will receive a financial reward for achieving monthly weight loss targets. Those who fail to meet their monthly goals will receive no financial reward. Such financial incentives have been considered in previous research. Due to the nature of the intervention, none of the investigative staff, trainers or subjects will be blinded to randomized assignment.

The primary objective of this study is to investigate whether a behavioral modification intervention in the form of either a 6-month supervised training program or a 6-month financial incentive program, results in overall superior clinical outcomes in comparison to standard of care. Specifically, improvement in glucose control, measured by A1c, will be considered. Given the objective nature of the Primary Outcome, there is little possibility of assessment bias of the primary or clinical outcomes.The secondary objective is to investigate the impact of a supervised training program and an incentivized weight loss program on weight-loss, LDL (apoB), blood pressure, waist-hip circumference, and diabetes-specific quality of life measures including behavioral and emotional impact (refer to Secondary Outcomes section).

Patients attending BCDiabetes ( Diabetes Clinic at Diamond Center )will be approached by one of their diabetes caregivers who will describe the study and determine whether they have interest in participating. If the patient expresses an interest, they will be provided additional information and a study consent form and be free to ask questions about the study. They may choose to provide consent at the time or to leave with the consent form and return at a later time to ask further questions. A research nurse, coordinator and/or co/principal investigator will be available to answer any questions the patient may have. When consent is provided, confirmation of the eligibility criteria will be completed and the subject will receive their randomized group assignment.

Eligible subjects will be randomized in a 2:1:1 fashion to the SoC, STP and IWL and groups respectively. Randomization will be stratified by age (≤ 50 vs > 50 years of age) to ensure balance in age groups in all three treatment arms; enrollment will not be stratified and the number of participants in the two age groups will not be restricted. Randomization within strata will be done in a permuted complete block design with random block sizes (blocks no smaller than 6 and no larger than 15). Randomization will be completed in advance and assignments will be kept in individual, separate sealed, sequentially labeled envelopes opened at the time of randomization of each individual.

Withdrawal from Study or Intervention:

Although they should be encouraged to continue participation in their randomized group, subjects can choose to withdraw from the study, or to withdraw from the intervention at any time. Subjects who choose to withdraw from the STP and IWL arms should continue to receive standard of care and will be considered cross-overs to SoC arm; these subjects are not necessarily withdrawing from the study and should be encouraged to continue to return for their scheduled 3 and 6 month study visits so study outcomes can be measured. If a subject chooses to withdraw from the study entirely, all attempts should be made to have them complete an exit visit where all study outcomes can be captured.

Subjects who experience any adverse event related to the STP arm (eg: physical injury while training) or experience the onset or worsening of an signs or symptoms related to a medical condition (eg: shortness of breath, dizziness, vomiting nausea, etc) persisting the day following a supervised training session, or who experience a worsening of a physical condition (eg: degenerative disc disorder, knee or hip pain, plantar fasciitis, etc) will be withdrawn from the STP intervention. As above, these subjects will be asked to return for their scheduled 3 and 6 month clinic visits.

If at any point more than 15% of subjects in the STP arm are withdrawn from the intervention arm due to an adverse event, worsening medical or physical condition, the study will be stopped.

Study data will be collected as part of the subject's electronic medical record at bcdiabetes.ca. Identifiable study data will be housed exclusively on bcdiabetes.ca; if removed from bcdiabetes.ca servers, subjects will be identified only with a study registration number different from their BC CareID number. Remote monitoring by EMMES using confidential authenticated automatically scheduled direct database queries. EMMES Canada will also provide oversight of quality assurance & monitoring.

The primary outcome measure is the percent of subjects who achieve target for A1c. The null and research hypothesis supporting the primary objective of investigating the impact of whether a behavioral modification intervention in the form of either a 6-month supervised training program or a 6-month incentivized weight loss program, results in overall superior clinical outcomes in comparison to standard of care is then:

H0: pSoC ≥ pIWL and pSoC ≥ pSTP vs. H1: pSoC < pIWL or pSoC < pSTP

where pSoC , pSTP and pIWL are the proportion of subjects achieving the target for all three disease measures. Here, rejecting the null hypothesis implies that the percent of patients achieving targets is higher in either of the STP arm or the IWL arm than in the SoC arm. A one-sided, 0.05 alpha-level simultaneous test for multiple contrasts of binomial proportions with an "Add-2" adjustment will be used.

The primary analysis cohort will be an ITT cohort including all randomized subjects and considering the arm to which they were originally randomized regardless of adherence to the regimen or the study protocol. Subjects who cross-over to the other intervention prior to Month 3 (ie: complete less than 3 of the required 6 months) will be considered failures in the arm to which they were originally randomized. Clinical data from the last, or exit visit will be used to construct the primary outcome for subjects who withdraw from the study, or from the intervention, subsequent to Month 3.

To corroborate the primary, unadjusted analysis, a logistic regression model will be fit with baseline clinical and demographic data as well as measures of compliance to intervention to adjust for possible imbalance of important variables. Also, the primary analysis will be repeated on a per-protocol cohort of subjects who completed the study according to the protocol and did not cross-over or withdraw from therapy. Graphical techniques and summary statistics for the two randomized groups at baseline and months 3 and 6 will also be presented.

Summary statistics and graphical presentations will be used to summarize data for all secondary outcomes. All hypothesis tests will be 2-sided and with a 5% Type I error probability. There will be no adjustment for multiple comparisons among the secondary outcomes with the exception that multiple domains within a single psychosocial instrument (eg: emotional burden, physician-related distress, regimen-related distress, and diabetes-related interpersonal distress domains within the DDS) will be subject to a Benjamini-Hochberg multiple comparison adjustment. Analyses will be conducted on the ITT cohort and corroborated by analysis on the per-protocol cohort.

Each clinical outcome measure is captured as a continuous and dichotomized variable (eg: A1c absolute level and those < 7.0%). Dichotomized variables will be analyzed as described in the Primary Analysis.

Continuous variables will be analyzed in three ways. First, summary statistics and graphical presentation of results will be performed for each of baseline and months 3 and 6. Second, change from baseline to month 6 will be compared using a paired t-test, or a Mann-Whitney test if distributional assumptions do not hold. A subject's last available, or exit visit, will be used if their month 6 visit is not available. Third, longitudinal random-effects models will be used to model the trajectory of each outcome over time and to determine the influence of randomized intervention group on that trajectory. Variables may be transformed to satisfy the assumptions of normally distributed random effects, but results will be presented on the original scale.

Sample Size Justification:

The primary null hypothesis compares the probability of a patient being in control in either experimental group to the Standard of Care group:

H0: pSoC ≥ pIWL and pSoC ≥ pSTP vs. H1: pSoC < pIWL or pSoC < pSTP

Based on data observed within the clinic from which cases are to be recruited, the success rate for Standard of Care patients is estimated to about 75%. A sample size of 200 subjects in a 2:1:1 randomization to the SoC, STP and IWL and groups respectively will provide a power of over 95% to reject the null hypothesis if the true difference between SoC and either experimental arm is 25% or greater (eg: 37.5% compared to 62.5%).

In addition, this sample size provides a power of more than 74% to reject the null hypothesis in favor of the alternative hypothesis that the percent of patients achieving control is greater among both the STP and IWL than among the SoC, if the true difference between arms is 25% or greater.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 or older.
2. Have been diagnosed with Type 2 diabetes by CDA guidelines.
3. A1c > 8.0 no more than 30 days prior to randomization and confirmed at the time of randomization.
4. Overweight or obese as defined by BMI of >25.

Exclusion Criteria:

1. Have medical co-morbidities that limit their exercise capacity (terminal cancer, severe physical disability such as limb amputation, blindness, seizure disorder, strokes with residual deficits, arrhythmias that would limit physical activity).
2. Alcohol or drug abuse that would interfere with exercise regimen.
3. Cannot read or write English (with the assistance of an interpreter) or are unable to fill out logs and questionnaire.
4. Inability or unwillingness of subject or legal guardian/representative to give written informed consent.
5. Patients for whom an exercise program is deemed medically inadvisable.
6. Patients already enrolled in a supervised training program.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2018-07 (Estimated); Primary Completion 2020-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Three months average blood glucose (A1c) | at 3 months and 6 months
  We will assess the effect of supervised training and financially incentivized weight loss on three month average blood glucose in patients with diabetes.

SECONDARY OUTCOMES:
apo B | 6 months
  proportion of patientst achieving apoB <0.8 mmol/L
systolic blood pressure (SBP) | 3 months and 6 months
  proportion of patients achieving SBP < 140 mmHg
A1c | 3 months and 6 months
  proportion of patients achieving A1c < 7.0%

OTHER OUTCOMES:
Composite: Psychosocial outcomes are depressive symptoms, Diabetes specific quality of life | 3 months and 6 months,
  this composite outcome will reflect overall change in QoL scoring during study
waist circumference | 3 months and 6 months,
  Waist circumference
weight | 3 months and 6 months,
  weight
body mass index (BMI) | 3 months and 6 months,
  BMI

CONTACTS AND LOCATIONS:
Overall Officials: Tom Elliott, MD, Principal Investigator — BCDiabetes.Ca
Locations (1):
- Vancouver General Hospital, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No
There is no plan to share IPD to other researchers except those involved in the trial

REFERENCES:
- [Background] Shaw JE, Sicree RA, Zimmet PZ. Global estimates of the prevalence of diabetes for 2010 and 2030. Diabetes Res Clin Pract. 2010 Jan;87(1):4-14. doi: 10.1016/j.diabres.2009.10.007. Epub 2009 Nov 6. PMID 19896746
- [Background] Klein S, Sheard NF, Pi-Sunyer X, Daly A, Wylie-Rosett J, Kulkarni K, Clark NG; American Diabetes Association; North American Association for the Study of Obesity; American Society for Clinical Nutrition. Weight management through lifestyle modification for the prevention and management of type 2 diabetes: rationale and strategies. A statement of the American Diabetes Association, the North American Association for the Study of Obesity, and the American Society for Clinical Nutrition. Am J Clin Nutr. 2004 Aug;80(2):257-63. doi: 10.1093/ajcn/80.2.257. PMID 15277143
- [Background] Anderson JW, Kendall CW, Jenkins DJ. Importance of weight management in type 2 diabetes: review with meta-analysis of clinical studies. J Am Coll Nutr. 2003 Oct;22(5):331-9. doi: 10.1080/07315724.2003.10719316. PMID 14559925